CLINICAL TRIAL: NCT06537557
Title: Application of an Early In-Hospital Temperature Management Protocol for Heat Stroke Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Jinhua Municipal Central Hospital (Other); Dongyang People's Hospital (Other); Lanxi People's Hospital (Other); Yiwu Central Hospital (Other); Jinhua People's Hospital (Unknown); Hangzhou Medical College (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0511
Record Dates: First submitted 2024-06-28; First posted 2024-08-05 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-06

CONDITIONS: Heat Stroke
MeSH Terms: conditions — Heat Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Using the early in-hospital temperature management protocol for heat stroke patients developed in our previous research, we will implement early identification, rapid cooling, and precise target temperature management for this group of patients.
  Interventions: Other: the early in-hospital temperature management protocol for heat stroke patients
- control group (No Intervention): We will retrospectively collect data on heat stroke patients who were visited before the implementation of the early in-hospital temperature management protocol between 2021 and 2022, meaning this group of patients received temperature management according to the original methods used by their respective hospitals.

INTERVENTIONS:
Other: the early in-hospital temperature management protocol for heat stroke patients — The early in-hospital temperature management protocol for heat stroke includes early identification, selection of cooling methods for rapid cooling, precise target temperature management, and dynamic monitoring. Effective temperature management will be implemented for heat stroke patients to improve their outcomes.
  Arms: experimental group

SUMMARY:
Heat stroke is a life-threatening clinical syndrome characterized by an imbalance between heat production and heat dissipation in the body, resulting from exposure to hot and humid environments and/or strenuous exercise. It is defined by an elevated core temperature exceeding 40°C and central nervous system abnormalities, accompanied by multi-organ dysfunction. The severity of cellular and tissue damage in heat stroke patients depends on the peak temperature reached and the duration of hyperthermia. Rapid reduction of core temperature can halt cellular damage, quickly reverse organ dysfunction, and improve patient outcomes. Therefore, early identification and rapid cooling are crucial to prevent irreversible damage and death in heat stroke patients. However, there is a lack of systematic and specific protocols to guide emergency medical staff in the standardized and effective management of body temperature in heat stroke patients. To address this, our research team previously developed an early in-hospital temperature management protocol for heat stroke patients based on the best available evidence, expert consultations, and expert panel meetings. This study aims to validate the feasibility and effectiveness of the protocol through clinical research, providing a basis for clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the emergency department and diagnosed with heat stroke according to the China expert consensus on Heat Stroke

Exclusion Criteria:

* transferred from another hospital and body temperature < 39.5℃; discharged within 4 hours, and subsequent body temperature or outcomes were unavailable; required immediate cardiopulmonary resuscitation; had other serious diseases, such as massive cerebral haemorrhage or severe trauma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
cooling rate at 0.5 hours | 0.5 hours
  The cooling rate at 0.5 hours was calculated in reference to initial body temperature and body temperature at 0.5 hours
Body temperature at 0.5 hours | 0.5 hours
  Body temperature at 0.5 hour refers to a reading obtained 25 to 35 minutes after admission.

SECONDARY OUTCOMES:
Body temperature at 2 hours | 2 hours
  Body temperature at 2 hours refers to a reading taken 100 to 140 minutes after admission
in-hospital mortality | 30 days
  Mortality from any cause during hospitalization
3-month mortality rate | 3 months
  death within 3 months after emergency visit
Number of participants with other complications | 3 months
  including heart failure, renal failure, coagulation disorders, respiratory failure, neurological sequelae, etc.

CONTACTS AND LOCATIONS:
Overall Officials: lan chen, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (7):
- China (7):
  - Yongkang First People's Hospital, Guli, Zhejiang
  - Dongyang People's Hospital, Dongyang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hanzhou
  - Jinhua Municipal Central Hospital, Jinhua
  - Jinhua People's Hospital, Jinhua
  - Lanxi People's Hospital, Lanxi
  - Yiwu Central Hospital, Yiwu